CLINICAL TRIAL: NCT07314801
Title: FINancial Toxicity and CAncer REcovery in YOUNG Adults
Acronym: FINCARE-Young
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Rami El Shafie, Prof. Dr., University Medical Center Goettingen
Other Study IDs: 20/7/25
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Financial Toxicity Related to Cancer Diagnosis and Tretment in Adolescents and Young Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and Young Adults with Cancer: This cohort consists of adolescents and young adults aged 18 to 39 years at the time of initial cancer diagnosis who received oncological treatment at a single tertiary care center. Participants have completed their primary cancer therapy and are assessed retrospectively and prospectively. The study does not involve any therapeutic intervention. Data are collected through structured telephone interviews and standardized questionnaires, complemented by clinical data extracted from electronic medical records. The focus of the cohort is to evaluate financial toxicity, socioeconomic factors, and employment-related outcomes following cancer treatment.

SUMMARY:
The FINCARE-Young study aims to investigate the extent and development of financial toxicity in adolescents and young adults with cancer. The primary purpose of this study is to assess the level of financial burden experienced during the acute phase of cancer treatment and after completion of therapy, and to analyze changes over time. In addition, the study seeks to identify sociodemographic, clinical, and socioeconomic factors associated with financial toxicity, as well as its impact on employment and social reintegration. By focusing on young adult cancer survivors, this study addresses an underexplored population and seeks to generate evidence to improve supportive care strategies and reduce long-term financial consequences of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 39 years at the time of initial cancer diagnosis
* Diagnosis of a malignant neoplasm
* Receipt of oncological treatment at the University Medical Center Göttingen
* Completion of primary cancer therapy at the time of study participation
* Initial diagnosis between 2014 and 2024
* Ability to provide informed consent
* Sufficient German language skills to participate in a telephone interview and complete questionnaires

Exclusion Criteria:

* Age below 18 years or above 39 years at the time of initial cancer diagnosis
* No history of malignant disease
* Ongoing primary cancer treatment at the time of study participation
* Severe cognitive impairment or psychiatric condition preventing reliable participation
* Insufficient German language proficiency to complete interviews or questionnaires
* Withdrawal of informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be selected from adolescents and young adults with a history of cancer who were treated at the University Medical Center Göttingen, a tertiary care academic hospital in Germany. Potential participants are identified through institutional clinical databases and electronic medical records. The source population includes individuals who received oncological care across all cancer entities within this center over the defined study period and who can be contacted for follow-up after completion of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Financial toxicity | From the acute phase of cancer treatment to the time of study participation after completion of therapy (retrospective assessment of treatment period and current assessment at follow-up), assessed only at one time point at study enrollment.
  Financial toxicity, assessed using the Comprehensive Score for Financial Toxicity (COST) questionnaire, measured during the acute phase of cancer treatment and at the time of study participation, including change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Rami El Shafie, Prof. Dr., Principal Investigator — University Medicine Göttingen
Locations (1):
- University Medicine Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves highly sensitive personal, medical, and socioeconomic information. Sharing individual-level data could pose a risk to participant privacy and confidentiality, even after pseudonymization, and is therefore not planned.